CLINICAL TRIAL: NCT02817880
Title: Comparison of the Analgesic Effect Between the Motor Cortex Stimulation (tDCS and rTMS) and the Trans-spinal Stimulation (tsDCS ) in the Algoneurodystrophy of Members. A Randomised Clinical Trial. tDCS : Transcranial Direct-current Stimulation rTMS : Repetitive Transcranial Magnetic Stimulation tsDCS : Transcutaneous Spinal Direct Current Stimulation
Brief Title: Comparison of the Analgesic Effect Between the Motor Cortex Stimulation and the Trans-spinal Stimulation in the Algoneurodystrophy.
Acronym: ALGOSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38RC15.158
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2022-05

CONDITIONS: Algoneurodystrophy
Keywords: rTMS, tDCS, tsDCS, pain, algoneurodystrophy , neurostimulation
MeSH Terms: conditions — Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- rTMS (repetitive transcranial magnetic stimulation) (Experimental): rTMS (repetitive transcranial magnetic stimulation)
  Interventions: Device: rTMS
- tDCS (transcranial direct-current stimulation) (Experimental): tDCS (transcranial direct-current stimulation)
  Interventions: Device: tDCS
- tsDCS (transcutaneous spinal Direct Current Stimulation) (Experimental): tsDCS (transcutaneous spinal Direct Current Stimulation)
  Interventions: Device: tsDCS

INTERVENTIONS:
Device: rTMS
  Arms: rTMS (repetitive transcranial magnetic stimulation)
Device: tDCS
  Arms: tDCS (transcranial direct-current stimulation)
Device: tsDCS
  Arms: tsDCS (transcutaneous spinal Direct Current Stimulation)

SUMMARY:
The purpose of this study is to compare the analgesic effectiveness of two motor cortex neurostimulations (tDCS and rTMS) and the trans-spinal neurostimulation (tsDCS ) in the algoneurodystrophy.

DETAILED DESCRIPTION:
* Entry into the study : After informed consent, patients will be randomised into three groups : tDCS, rTMS, tsDCS. The physician responsible for conducting neurostimulation sessions will make the randomization via an interactive web response system (IWRS).
* Baseline : Participants, will record on a book, a daily Visual Numeric Scale(VNS) of Pain Intensity for 1 month.
* The beginning of the treatment : after the baseline, sessions of neurostimulation will begin. Sessions of neurostimulation will have a decreasing rhythm. Five sessions per week during the two first weeks, two sessions per week during the third week, one session during the fourth week and then two sessions per month for four months.
* After the end of neurostimulation sessions, patients will be followed for 1month.

Throughout their participation in the study, patients will complete their VNS report book (1month of baseline before the treatment, 3 months during neurostimulation, 1 month after neurostimulation).

Patients will have 5 evaluation examinations:

* The first, one just before the beginning of the neurostimulation,
* The second, 1 month after the beginning of neurostimulation
* The third, 3 months after the beginning of neurostimulation
* And the last one, 1 month after the end of neurostimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patient's written consent
* Patient suffering from an algoneurodystrophy for more than a year.
* Diagnosis of algoneurodystrophy confirmed by an osseous scintigraphy
* Stable treatment for at least 1 month
* Patient non-responsive to pharmacological treatments
* VNS > 3 at the time of screening

Exclusion Criteria:

* Drug addiction
* History of epilepsy, head trauma, Psychiatric pathology likely to hamper the progress of the study.
* Intracranial ferromagnetic material or an implanted stimulator
* MRI contraindication
* Algoneurodystrophy due to a nervous lesion
* Pregnant women, parturient women, breast-feeding mother. Lack of effective contraception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
The Visual numeric scale of pain between the three groups | Baseline to 1 month

SECONDARY OUTCOMES:
The Clinical Global Impression scale (CGI) between the three groups | Baseline, 3 months after the beginning of the treatment (day 90), and 1 month after the end of the treatment (Day 180)
The SF12 quality of life questionnaire between the three groups | Baseline, 3 months after the beginning of the treatment (day 90), and 1 month after the end of the treatment (Day 180)
The Hospital Anxiety and Depression scale (HAD) between the three groups | Baseline, 3 months after the beginning of the treatment (day 90), and 1 month after the end of the treatment (Day 180)
The Neuropathic Pain Symptom Inventory scale (NPSI) between the three groups | Baseline, 3 months after the beginning of the treatment (day 90), and 1 month after the end of the treatment (Day 180)
Evolution of the conductance of feet and hands by using Sudoscan | Baseline, 3 months after the beginning of the treatment (day 90), and 1 month after the end of the treatment (Day 180)
  The body conductance will be used to assess the evolution of the Impact of the neurostimulation on the sympathetic nervous system and on the small fiber neuropathy.
Modifications of the sensori-motor cortical cards by using a MRI | Baseline, and 1 month after the end of the treatment (Day 180)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre de la douleur, CHU Grenoble Alpes, Grenoble, Isere
  - Service de Physiologie - Explorations Fonctionnelles, Hôpital Henri Mondor, Créteil, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lefaucheur JP, Drouot X, Menard-Lefaucheur I, Keravel Y, Nguyen JP. Motor cortex rTMS restores defective intracortical inhibition in chronic neuropathic pain. Neurology. 2006 Nov 14;67(9):1568-74. doi: 10.1212/01.wnl.0000242731.10074.3c. PMID 17101886
- [Background] de Andrade DC, Mhalla A, Adam F, Texeira MJ, Bouhassira D. Neuropharmacological basis of rTMS-induced analgesia: the role of endogenous opioids. Pain. 2011 Feb;152(2):320-326. doi: 10.1016/j.pain.2010.10.032. Epub 2010 Dec 10. PMID 21146300
- [Background] Lefaucheur JP, Andre-Obadia N, Poulet E, Devanne H, Haffen E, Londero A, Cretin B, Leroi AM, Radtchenko A, Saba G, Thai-Van H, Litre CF, Vercueil L, Bouhassira D, Ayache SS, Farhat WH, Zouari HG, Mylius V, Nicolier M, Garcia-Larrea L. [French guidelines on the use of repetitive transcranial magnetic stimulation (rTMS): safety and therapeutic indications]. Neurophysiol Clin. 2011 Dec;41(5-6):221-95. doi: 10.1016/j.neucli.2011.10.062. Epub 2011 Nov 10. French. PMID 22153574
- [Background] Lefaucheur JP, Menard-Lefaucheur I, Goujon C, Keravel Y, Nguyen JP. Predictive value of rTMS in the identification of responders to epidural motor cortex stimulation therapy for pain. J Pain. 2011 Oct;12(10):1102-11. doi: 10.1016/j.jpain.2011.05.004. Epub 2011 Jul 31. PMID 21807565
- [Background] Lefaucheur, J. P. (2007).
- [Background] Khedr EM, Kotb H, Kamel NF, Ahmed MA, Sadek R, Rothwell JC. Longlasting antalgic effects of daily sessions of repetitive transcranial magnetic stimulation in central and peripheral neuropathic pain. J Neurol Neurosurg Psychiatry. 2005 Jun;76(6):833-8. doi: 10.1136/jnnp.2004.055806. PMID 15897507
- [Background] Passard A, Attal N, Benadhira R, Brasseur L, Saba G, Sichere P, Perrot S, Januel D, Bouhassira D. Effects of unilateral repetitive transcranial magnetic stimulation of the motor cortex on chronic widespread pain in fibromyalgia. Brain. 2007 Oct;130(Pt 10):2661-70. doi: 10.1093/brain/awm189. Epub 2007 Sep 14. PMID 17872930
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Leung A, Donohue M, Xu R, Lee R, Lefaucheur JP, Khedr EM, Saitoh Y, Andre-Obadia N, Rollnik J, Wallace M, Chen R. rTMS for suppressing neuropathic pain: a meta-analysis. J Pain. 2009 Dec;10(12):1205-16. doi: 10.1016/j.jpain.2009.03.010. Epub 2009 May 23. PMID 19464959
- [Background] Lefaucheur JP. Use of repetitive transcranial magnetic stimulation in pain relief. Expert Rev Neurother. 2008 May;8(5):799-808. doi: 10.1586/14737175.8.5.799. PMID 18457536
- [Background] Nitsche MA, Liebetanz D, Lang N, Antal A, Tergau F, Paulus W. Safety criteria for transcranial direct current stimulation (tDCS) in humans. Clin Neurophysiol. 2003 Nov;114(11):2220-2; author reply 2222-3. doi: 10.1016/s1388-2457(03)00235-9. No abstract available. PMID 14580622
- [Background] Nitsche MA, Paulus W. Sustained excitability elevations induced by transcranial DC motor cortex stimulation in humans. Neurology. 2001 Nov 27;57(10):1899-901. doi: 10.1212/wnl.57.10.1899. PMID 11723286
- [Background] Medeiros LF, de Souza IC, Vidor LP, de Souza A, Deitos A, Volz MS, Fregni F, Caumo W, Torres IL. Neurobiological effects of transcranial direct current stimulation: a review. Front Psychiatry. 2012 Dec 28;3:110. doi: 10.3389/fpsyt.2012.00110. eCollection 2012. PMID 23293607
- [Background] Thibaut A, Chatelle C, Gosseries O, Laureys S, Bruno MA. [Transcranial direct current stimulation: a new tool for neurostimulation]. Rev Neurol (Paris). 2013 Feb;169(2):108-20. doi: 10.1016/j.neurol.2012.05.008. Epub 2012 Sep 7. French. PMID 22959705
- [Background] Fregni F, Gimenes R, Valle AC, Ferreira MJ, Rocha RR, Natalle L, Bravo R, Rigonatti SP, Freedman SD, Nitsche MA, Pascual-Leone A, Boggio PS. A randomized, sham-controlled, proof of principle study of transcranial direct current stimulation for the treatment of pain in fibromyalgia. Arthritis Rheum. 2006 Dec;54(12):3988-98. doi: 10.1002/art.22195. PMID 17133529
- [Background] Antal A, Kriener N, Lang N, Boros K, Paulus W. Cathodal transcranial direct current stimulation of the visual cortex in the prophylactic treatment of migraine. Cephalalgia. 2011 May;31(7):820-8. doi: 10.1177/0333102411399349. Epub 2011 Mar 11. PMID 21398419
- [Background] Fregni F, Boggio PS, Lima MC, Ferreira MJ, Wagner T, Rigonatti SP, Castro AW, Souza DR, Riberto M, Freedman SD, Nitsche MA, Pascual-Leone A. A sham-controlled, phase II trial of transcranial direct current stimulation for the treatment of central pain in traumatic spinal cord injury. Pain. 2006 May;122(1-2):197-209. doi: 10.1016/j.pain.2006.02.023. Epub 2006 Mar 27. PMID 16564618
- [Background] Mori F, Codeca C, Kusayanagi H, Monteleone F, Buttari F, Fiore S, Bernardi G, Koch G, Centonze D. Effects of anodal transcranial direct current stimulation on chronic neuropathic pain in patients with multiple sclerosis. J Pain. 2010 May;11(5):436-42. doi: 10.1016/j.jpain.2009.08.011. Epub 2009 Dec 16. PMID 20018567
- [Background] Antal A, Terney D, Kuhnl S, Paulus W. Anodal transcranial direct current stimulation of the motor cortex ameliorates chronic pain and reduces short intracortical inhibition. J Pain Symptom Manage. 2010 May;39(5):890-903. doi: 10.1016/j.jpainsymman.2009.09.023. PMID 20471549
- [Background] O'Connell NE, Wand BM, Marston L, Spencer S, Desouza LH. Non-invasive brain stimulation techniques for chronic pain. A report of a Cochrane systematic review and meta-analysis. Eur J Phys Rehabil Med. 2011 Jun;47(2):309-26. Epub 2011 Apr 14. PMID 21494222
- [Background] Zaghi S, Thiele B, Pimentel D, Pimentel T, Fregni F. Assessment and treatment of pain with non-invasive cortical stimulation. Restor Neurol Neurosci. 2011;29(6):439-51. doi: 10.3233/RNN-2011-0615. PMID 22124038
- [Background] Luedtke K, Rushton A, Wright C, Geiss B, Juergens TP, May A. Transcranial direct current stimulation for the reduction of clinical and experimentally induced pain: a systematic review and meta-analysis. Clin J Pain. 2012 Jun;28(5):452-61. doi: 10.1097/AJP.0b013e31823853e3. PMID 22569218
- [Background] O'Connell NE, Wand BM, Marston L, Spencer S, Desouza LH. Non-invasive brain stimulation techniques for chronic pain. Cochrane Database Syst Rev. 2014 Apr 11;(4):CD008208. doi: 10.1002/14651858.CD008208.pub3. PMID 24729198
- [Background] Cogiamanian F, Vergari M, Pulecchi F, Marceglia S, Priori A. Effect of spinal transcutaneous direct current stimulation on somatosensory evoked potentials in humans. Clin Neurophysiol. 2008 Nov;119(11):2636-40. doi: 10.1016/j.clinph.2008.07.249. Epub 2008 Sep 10. PMID 18786856
- [Background] Truini A, Vergari M, Biasiotta A, La Cesa S, Gabriele M, Di Stefano G, Cambieri C, Cruccu G, Inghilleri M, Priori A. Transcutaneous spinal direct current stimulation inhibits nociceptive spinal pathway conduction and increases pain tolerance in humans. Eur J Pain. 2011 Nov;15(10):1023-7. doi: 10.1016/j.ejpain.2011.04.009. Epub 2011 May 14. PMID 21576030
- [Background] Toshev PK, Guleyupoglu B, Bikson M. Informing dose design by modeling transcutaneous spinal direct current stimulation. Clin Neurophysiol. 2014 Nov;125(11):2147-2149. doi: 10.1016/j.clinph.2014.03.022. Epub 2014 Apr 4. No abstract available. PMID 24775922
- [Background] Priori A, Ciocca M, Parazzini M, Vergari M, Ferrucci R. Transcranial cerebellar direct current stimulation and transcutaneous spinal cord direct current stimulation as innovative tools for neuroscientists. J Physiol. 2014 Aug 15;592(16):3345-69. doi: 10.1113/jphysiol.2013.270280. Epub 2014 Jun 6. PMID 24907311
- [Background] Cogiamanian F, Ardolino G, Vergari M, Ferrucci R, Ciocca M, Scelzo E, Barbieri S, Priori A. Transcutaneous spinal direct current stimulation. Front Psychiatry. 2012 Jul 4;3:63. doi: 10.3389/fpsyt.2012.00063. eCollection 2012. PMID 22783208
- [Background] Plow EB, Pascual-Leone A, Machado A. Brain stimulation in the treatment of chronic neuropathic and non-cancerous pain. J Pain. 2012 May;13(5):411-24. doi: 10.1016/j.jpain.2012.02.001. Epub 2012 Apr 7. PMID 22484179
- [Background] Lefaucheur JP, Antal A, Ahdab R, Ciampi de Andrade D, Fregni F, Khedr EM, Nitsche M, Paulus W. The use of repetitive transcranial magnetic stimulation (rTMS) and transcranial direct current stimulation (tDCS) to relieve pain. Brain Stimul. 2008 Oct;1(4):337-44. doi: 10.1016/j.brs.2008.07.003. Epub 2008 Oct 7. PMID 20633392
- [Background] Fregni F, Freedman S, Pascual-Leone A. Recent advances in the treatment of chronic pain with non-invasive brain stimulation techniques. Lancet Neurol. 2007 Feb;6(2):188-91. doi: 10.1016/S1474-4422(07)70032-7. PMID 17239806
- [Background] Nizard J, Lefaucheur JP, Helbert M, de Chauvigny E, Nguyen JP. Non-invasive stimulation therapies for the treatment of refractory pain. Discov Med. 2012 Jul;14(74):21-31. PMID 22846200
- [Background] Mhalla A, Baudic S, de Andrade DC, Gautron M, Perrot S, Teixeira MJ, Attal N, Bouhassira D. Long-term maintenance of the analgesic effects of transcranial magnetic stimulation in fibromyalgia. Pain. 2011 Jul;152(7):1478-1485. doi: 10.1016/j.pain.2011.01.034. Epub 2011 Mar 11. PMID 21397400
- [Background] Zaghi S, DaSilva AF, Acar M, Lopes M, Fregni F. One-year rTMS treatment for refractory trigeminal neuralgia. J Pain Symptom Manage. 2009 Oct;38(4):e1-5. doi: 10.1016/j.jpainsymman.2009.04.020. Epub 2009 Aug 26. No abstract available. PMID 19713068
- [Background] Lefaucheur JP, Drouot X, Menard-Lefaucheur I, Nguyen JP. Neuropathic pain controlled for more than a year by monthly sessions of repetitive transcranial magnetic stimulation of the motor cortex. Neurophysiol Clin. 2004 Apr;34(2):91-5. doi: 10.1016/j.neucli.2004.02.001. PMID 15130555
- [Background] Hodaj H, Alibeu JP, Payen JF, Lefaucheur JP. Treatment of Chronic Facial Pain Including Cluster Headache by Repetitive Transcranial Magnetic Stimulation of the Motor Cortex With Maintenance Sessions: A Naturalistic Study. Brain Stimul. 2015 Jul-Aug;8(4):801-7. doi: 10.1016/j.brs.2015.01.416. Epub 2015 Feb 7. PMID 25979838
- [Background] Kim YJ, Ku J, Kim HJ, Im DJ, Lee HS, Han KA, Kang YJ. Randomized, sham controlled trial of transcranial direct current stimulation for painful diabetic polyneuropathy. Ann Rehabil Med. 2013 Dec;37(6):766-76. doi: 10.5535/arm.2013.37.6.766. Epub 2013 Dec 23. PMID 24466511
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Picarelli H, Teixeira MJ, de Andrade DC, Myczkowski ML, Luvisotto TB, Yeng LT, Fonoff ET, Pridmore S, Marcolin MA. Repetitive transcranial magnetic stimulation is efficacious as an add-on to pharmacological therapy in complex regional pain syndrome (CRPS) type I. J Pain. 2010 Nov;11(11):1203-10. doi: 10.1016/j.jpain.2010.02.006. Epub 2010 Apr 28. PMID 20430702
- [Background] M. Sorel, J.-P. Lefaucheur, J.-C. Beatrix, A.M. Domec, M.L. Giboutet, E. Houy, J. Robert, P. Cesaro (2012); Complex regional pain syndrome: interest in coupling the vascular phase of technetium 99 bone scintigraphy with the effectiveness of ketamine. Lett. Méd. Phys. Réadapt., OI 10.1007/s11659-012-0296-1
- [Result] Delon-Martin C, Lefaucheur JP, Hodaj E, Sorel M, Dumolard A, Payen JF, Hodaj H. Neural Correlates of Pain-Autonomic Coupling in Patients With Complex Regional Pain Syndrome Treated by Repetitive Transcranial Magnetic Stimulation of the Motor Cortex. Neuromodulation. 2024 Jan;27(1):188-199. doi: 10.1016/j.neurom.2023.05.005. Epub 2023 Aug 16. PMID 37589642
- [Result] Lefaucheur JP, Delon-Martin C, Hodaj H. Functional coupling between chronic pain and the autonomic nervous system revealed by neuromodulation techniques. Comment on 'Effect of neuromodulation for chronic pain on the autonomic nervous system: a systematic review' (BJA Open 2024; 11: 100305). BJA Open. 2025 Mar 29;14:100393. doi: 10.1016/j.bjao.2025.100393. eCollection 2025 Jun. No abstract available. PMID 40223918
- [Result] Hodaj H, Payen JF, Hodaj E, Sorel M, Dumolard A, Vercueil L, Delon-Martin C, Lefaucheur JP. Long-term analgesic effect of trans-spinal direct current stimulation compared to non-invasive motor cortex stimulation in complex regional pain syndrome. Brain Commun. 2023 Jul 1;5(4):fcad191. doi: 10.1093/braincomms/fcad191. eCollection 2023. PMID 37545548